CLINICAL TRIAL: NCT04106726
Title: A MULTI-CENTER, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, PARALLEL-GROUP STUDY, COMPARING IVERMECTIN CREAM 1% (ZYDUS WORLDWIDE DMCC) TO SOOLANTRA® (GALDERMA LABORATORIES, L.P.) AND BOTH ACTIVE TREATMENTS TO A PLACEBO CONTROL IN THE TREATMENT OF MODERATE TO SEVERE FACIAL ROSACEA
Brief Title: Bioequivalence Study of Ivermectin Cream 1% in Treatment of Moderate to Severe Facial Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zydus Worldwide DMCC (Industry)
Collaborators: Catawba Research, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVRC 1907
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Facial Rosacea
Keywords: Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test: Ivermectin cream 1% (Experimental): Manufactured by Zydus Worldwide DMCC; Apply cream to the affected areas of the face once daily for 12 weeks.
  Interventions: Drug: Ivermectin cream 1%
- Reference: Soolantra® cream, 1% (Active Comparator): Manufactured by Galderma Laboratories, L.P.; Apply cream to the affected areas of the face once daily for 12 weeks.
  Interventions: Drug: Soolantra® Ivermectin cream 1%
- Placebo: Placebo for Ivermectin cream 1% (Placebo Comparator): Manufactured by Zydus Worldwide DMCC; Apply to the affected areas of the face once daily for 12 weeks.
  Interventions: Drug: Placebo for Ivermectin cream 1%

INTERVENTIONS:
Drug: Soolantra® Ivermectin cream 1% — Apply topically to the face once daily for 84 consecutive days.
  Arms: Reference: Soolantra® cream, 1%
Drug: Ivermectin cream 1% — Apply topically to the face once daily for 84 consecutive days.
  Arms: Test: Ivermectin cream 1%
Drug: Placebo for Ivermectin cream 1% — Apply topically to the face once daily for 84 consecutive days.
  Arms: Placebo: Placebo for Ivermectin cream 1%

SUMMARY:
To evaluate the therapeutic equivalence and safety of ivermectin cream 1% (Zydus Worldwide DMCC) and Soolantra® (ivermectin) cream, 1% (Galderma Laboratories, L.P.) in the treatment of moderate to severe facial papulopustular rosacea.

To demonstrate the superiority of the efficacy of the test and reference products over that of the placebo control in the treatment of moderate to severe facial rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female aged ≥ 18 years with a clinical diagnosis of facial papulopustular rosacea.
2. Subjects must have provided IRB approved written informed consent.
3. Subjects must have at least 15 and not more than 50 inflammatory facial lesions (i.e., papules/pustules) at screening and baseline visits. For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area including those present on the nose. Lesions involving the eyes, and scalp will be excluded from the count.
4. Subjects must have no more than 2 nodulocystic lesions on the face at Screening and Baseline visits.
5. Subjects must have a definite clinical diagnosis of facial papulopustular rosacea severity grade 3 or 4 as per the Investigator Global Assessment (IGA) (per Table 1 below) at screening and baseline visits.
6. Subjects must have persistent erythema on the face with moderate (2) score or higher (per table 2 below) at screening and baseline visits.
7. Subjects must have a mild (1) to moderate (2) score for telangiectasia on the face. (per table 3 below) at screening and baseline visits.
8. 8. Subjects must be willing to minimize external factors that might trigger rosacea flare-ups (e.g., spicy foods, thermally hot foods and drinks, hot environments, prolonged sun exposure, strong winds and alcoholic beverages)
9. Subjects must be willing to refrain from using all other topical medications for rosacea during the 12-week treatment period, other than the investigational product.
10. Female Subjects of childbearing potential (excluding women who are or premenarchal, surgically sterilized (by hysterectomy) or postmenopausal for at least 1 year prior to screening), in addition to having a negative urine pregnancy test, must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to 30 days after the last administration of study drug. For the purpose of this study the following are considered acceptable methods of birth control: oral or injectable contraceptives, contraceptive patches, Depo-Provera® (stabilized for at least 3 months prior to screening), NuvaRing® (vaginal contraceptive), Implanon™ (contraceptive implant), double-barrier methods (e.g. condom and spermicide), IUD, or abstinence with a 2nd acceptable method of birth control should the Subject become sexually active. Subjects on hormonal contraception must be stabilized on the same type for at least three months prior to screening and must not change the method during the study. A sterile sexual partner is NOT considered an adequate form of birth control.
11. All male Subjects must agree to use accepted methods of birth control with their partners, from the day of the first dose administration to 30 days after the last administration of study drug. Abstinence is an acceptable method of birth control. Female partners should use an acceptable method of birth control as described in the above Item Number 10.
12. Subjects who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to screening and must agree to not change make-up brand/type or frequency of use throughout the study.
13. Subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits.
14. Subjects must be in good health and free from any clinically significant disease, including but not limited to, conditions that may interfere with the evaluation of facial rosacea. Such conditions include but are not limited to the following: autoimmune disease; acne vulgaris on the face; seborrheic dermatitis on the face; perioral dermatitis; corticosteroid-induced acne; carcinoid syndrome; mastocytosis; acneiform eruptions caused by make-up, medication, facial psoriasis and facial eczema.

Exclusion Criteria:

1. Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
2. Subjects with a history of hypersensitivity or allergy to ivermectin, propylene glycol and/or any of the study medication ingredients and its excipients.
3. Subjects with the presence of other forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other dermatoses that may be confounded with papulopustular rosacea, such as peri-oral dermatitis, facial keratosis pilaris, seborrheic dermatitis and acne.
4. Subjects with excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of facial rosacea.
5. Subjects with moderate or severe rhinophyma, dense telangiectases (score 3, severe), or plaque-like facial edema.
6. Subjects with a severe irritation (score 3 = severe (marked/intense)) for dryness, pruritus, or stinging/burning.
7. Subjects with ocular rosacea (e.g., conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.
8. Subjects who currently have or have recently had bacterial folliculitis on the face.
9. Subjects who have unstable medical disorders that are clinically significant or have lifethreatening diseases. Subjects who have clinically significant abnormal laboratory values according to the investigator at screening.
10. Subjects who had within 14 days prior to screening:

    1. wax depilation of the face
    2. cosmetic procedures (e.g., facials) which may affect assessment of facial rosacea
    3. exposure to excessive UV radiation or the subject is planning exposure during the study (e.g. occupational exposure to the sun, planned holidays in the sun during the study, phototherapy, tanning salon),
    4. used a sauna.
11. Subjects who have used any of the following procedures on the face within 1 month prior to screening:

    1. cryodestruction or chemodestruction,
    2. dermabrasion,
    3. photodynamic therapy,
    4. acne surgery,
    5. intralesional steroids, or
    6. X-ray therapy.
12. Subjects who have used any of the following topical treatments on the face within 1 month prior to screening:

    1. retinoids
    2. benzoyl peroxide
    3. immunomodulators
    4. antibiotics (e.g., metronidazole and macrolides)
    5. corticosteroids
    6. other topical rosacea treatment (e.g., azelaic acid, metronidazole) or topical erythema treatment (e.g. brimonidine)
13. Subjects who have used any of the following systemic treatments within 1 month prior to screening:

    1. corticosteroids,
    2. systemic antibiotics known to have an impact on the severity of facial rosacea (e.g., containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim),
    3. other systemic treatments that affect erythema: alpha-blockers (e.g., mirtazapine), beta-blockers (e.g., propranolol), alpha 2 agonist (e.g., clonidine), or
    4. other systemic treatment for rosacea.
14. Subjects who have used any of the following topical treatments within 6 weeks prior to screening:

    1. corticosteroids,
    2. antibiotics for rosacea,
    3. medications for rosacea (e.g., azelaic acid, metronidazole),
    4. over-the-counter preparations for rosacea, or
    5. anti-inflammatory agents. Note: Non-steroidal anti-inflammatory drugs (NSAIDs) and aspirin use on an as needed basis and if not used consecutively for > 14 days prior to screening and/or during the study is acceptable. Note: Low dose (81 mg) aspirin taken daily is acceptable.
15. Subjects who have used or changed their use of estrogens or oral contraceptives within the 3 months prior to screening.
16. Subjects who have received radiation therapy and/or anti-neoplastic agents within 3 months prior to screening.
17. Subjects who have used within 6 months prior to screening antiandrogens such as Spironolactone, oral retinoids (e.g. Accutane®), or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
18. Subjects who have had laser therapy (for telangiectasia or other conditions), electrodessication and phototherapy (e.g., ClearLight®) to the facial area within 6 months prior to study entry (Visit 1 Screening Visit).
19. Subjects who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold.
20. Subjects who consume excessive amounts of alcohol (greater than two drinks per day) or use drugs of abuse (including, but not limited to, cannabinoids, cocaine and barbiturates).
21. Subjects who have participated in an investigational drug study (i.e., Subjects have been treated with an investigational drug) within 30 days prior to screening will be excluded from study participation. Subjects who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion.
22. Subjects who have been previously enrolled in this study.
23. Subjects who live in the same household with subjects currently enrolled in this trial.
24. Subjects who have a history of being unresponsive to topical ivermectin therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Mean percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts. | 12 weeks
  Mean percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts.

SECONDARY OUTCOMES:
Exploratory Endpoint: The proportion of subjects with a clinical response (IGA) of "success" at week 12. | 12 weeks
  The proportion of subjects with a clinical response (IGA) of "success" at week 12.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Zydus Worldwide DMCC, Brandon, Florida
  - Zydus Worldwide DMCC, Fort Lauderdale, Florida
  - Zydus Worldwide DMCC, Miami, Florida
  - Zydus Worldwide DMCC, Miramar, Florida
  - Zydus Worldwide DMCC, Tampa, Florida
  - Zydus Worldwide DMCC, Saginaw, Michigan
  - Zydus Worldwide DMCC, High Point, North Carolina
  - Zydus Worldwide DMCC, Sugarloaf, Pennsylvania
  - Zydus Worldwide DMCC, Upper Saint Clair, Pennsylvania
  - Zydus Worldwide DMCC, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No